CLINICAL TRIAL: NCT05162482
Title: Immunogenicity and Safety of Heterologous Combinations of COVID-19 Vaccines Available Under Emergency Use Authorization in Pakistan: A Randomized Phase II Trial
Brief Title: Combination Assessment Trial of COVID-19 Vaccines (COMBAT-COVID)
Acronym: COMBAT-COVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); University of Oxford (Other); International Vaccine Institute (Other); Harvard Medical School (HMS and HSDM) (Other); Chughtai Lab (Unknown); National Institute of Health, Pakistan (Unknown)
Responsible Party: Principal Investigator, Dr. Farah Qamar, Associate Professor, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6739
Record Dates: First submitted 2021-12-13; First posted 2021-12-17 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: COVID 19 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Heterologous 1 (Active Comparator): BIBP (CNBG, Sinopharm) WIV (0.5ml) at baseline CanSinoBIO (0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: BIBP (CNBG, Sinopharm) WIV; Biological: CanSinoBIO
- Heterologous 2 (Active Comparator): BIBP (CNBG, Sinopharm) WIV (0.5ml) at baseline AstraZeneca ChAdOx (0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: BIBP (CNBG, Sinopharm) WIV; Biological: AstraZeneca ChAdOx
- Heterologous 3 (Active Comparator): CanSinoBIO (0.5ml) at baseline BIBP (CNBG, Sinopharm) WIV (0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: BIBP (CNBG, Sinopharm) WIV; Biological: CanSinoBIO
- Heterologous 4 (Active Comparator): CanSinoBIO (0.5ml) at baseline AstraZeneca ChAdOx (0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: CanSinoBIO; Biological: AstraZeneca ChAdOx
- Heterologous 5 (Active Comparator): AstraZeneca ChAdOx (0.5ml) at baseline BIBP (CNBG, Sinopharm) WIV(0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: BIBP (CNBG, Sinopharm) WIV; Biological: AstraZeneca ChAdOx
- Heterologous 6 (Active Comparator): AstraZeneca ChAdOx (0.5ml) at baseline CanSinoBIO (0.5ml) after 70±7 days (10 wks±2)
  (160 participants)
  Interventions: Biological: CanSinoBIO; Biological: AstraZeneca ChAdOx
- Homologous 7 (Active Comparator): BIBP (CNBG, Sinopharm) WIV (0.5ml) at baseline BIBP (CNBG, Sinopharm) WIV (0.5ml) after 70±7 days (10 wks±2) Full dose booster: 80 participants (0.5ml) 6 months after second dose Fractional dose booster: 80 participants (dose to be decided) 6 months after second dose No booster: 80 participants
  (240 participants)
  Interventions: Biological: BIBP (CNBG, Sinopharm) WIV
- Homologous 8 (Active Comparator): CanSinoBIO (0.5ml) at baseline CanSinoBIO (0.5ml) after 70±7 days (10 wks±2) Full dose booster: 80 participants (0.5ml) 6 months after second dose Fractional dose booster: 80 participants (dose to be decided) 6 months after second dose No booster: 80 participants
  (240 participants)
  Interventions: Biological: CanSinoBIO
- Homologous 9 (Active Comparator): AstraZeneca ChAdOx (0.5ml) at baseline AstraZeneca ChAdOx (0.5ml) after 70±7 days (10 wks±2) Full dose booster: 80 participants (0.5ml) 6 months after second dose Fractional dose booster: 80 participants (dose to be decided) 6 months after second dose No booster: 80 participants
  (240 participants)
  Interventions: Biological: AstraZeneca ChAdOx

INTERVENTIONS:
Biological: BIBP (CNBG, Sinopharm) WIV — BIBP (CNBG, Sinopharm) WIV (Whole Inactivated Virus in a single dose, prefilled syringe with a storage temperature of 2-8°C)
  Arms: Heterologous 1; Heterologous 2; Heterologous 3; Heterologous 5; Homologous 7
Biological: CanSinoBIO — CanSinoBIO (Viral Vector in a single dose, prefilled syringe with a storage temperature of 2-8°C)
  Arms: Heterologous 1; Heterologous 3; Heterologous 4; Heterologous 6; Homologous 8
Biological: AstraZeneca ChAdOx — AstraZeneca ChAdOx (Viral Vector in a multi-dose vial consisting of 10 doses with a storage temperature of 2-8°C)
  Arms: Heterologous 2; Heterologous 4; Heterologous 5; Heterologous 6; Homologous 9

SUMMARY:
This is a randomized, phase II trial which will be conducted among volunteers aged 18 years and above in Karachi, Lahore and Islamabad, Pakistan. The trial will have nine arms and is an open label study. Trained persons will administer the vaccine and draw blood under strict aseptic measures. The immune responses using pseudo neutralizing antibodies against SARS-CoV-2 in COVID-19 seronegative participants receiving heterologous and homologous COVID-19 vaccines will be assessed. Anti-spike IgG antibodies by ELISA and pseudo neutralizing antibodies against SARS-CoV-2 will also be measured. The safety and reactogenicity will also be assessed by recording serious adverse events (SAE), adverse events of special interest (AESI), solicited local and systemic reactions and medically attended adverse reactions through biochemical and hematological tests or safety measures throughout the study. In most cases the adverse events are mild and self-limiting but can require medication and/or hospitalization in rare cases. Participants suffering from any adverse event causally related to the to the trial intervention will be facilitated and the cost of treatment including laboratory investigations will be provided to them. Data confidentiality will be ensured by delinking names in forms and through password protection.

DETAILED DESCRIPTION:
This is a randomized, phase II trial which will be conducted among volunteers aged 18 years and above in Karachi, Lahore and Islamabad, Pakistan. The investigators will be assessing the safety and reactogenicity of heterologous and homologous COVID-19 vaccines and characterize the immune responses using pseudo neutralizing antibodies against SARS-CoV-2 in COVID seronegative participants immunized with heterologous and homologous COVID-19 vaccines regimens. This approach will allow combination of different vaccines in case the same vaccine is not available at the time of boosting (follow-up dose) and will help mitigate the shortage of available COVID-19 vaccines. Furthermore, the combination strategy might prove to be more effective against the variants of concern of SARS CoV-2.

The total duration of the trial will be approximately 2 ½ years. The study will enroll participants which will be divided into 2 cohorts, one for a more detailed immunological assessment and one for main immunology endpoints. The study will include 9 study groups with different combinations of COVID-19 vaccine schedule (6 heterologous combinations and 3 homologous combinations plus booster in homologous arms). The investigators will be measuring Anti-spike IgG antibodies by ELISA at week 14 (4 weeks post booster dose) and pseudo neutralizing antibodies against SARS-CoV-2 at day 0, and weeks 4, 14, 24, 28, 48, 60 and 96 as per schedule of events for the immunology cohort and at baseline and 4 weeks post second dose in general cohort. This is a pragmatic trial where the interval between the two doses will be kept longer than the conventional recommendations of 21/28 days. Additionally, the investigators will also be assessing safety and reactogenicity by recording serious adverse events (SAE), adverse events of special interest (AESI), solicited local and systemic reactions within 7 days post each dose, unsolicited reactions within 28 days post each dose, medically attended adverse reactions up to 3 months post booster dose and changes from baseline to 4 weeks post each dose in biochemical and hematological tests or safety measures throughout the study.

A trained person will administer the vaccine and draw blood samples under strict aseptic techniques to ensure minimum discomfort and reduce the risk of infection. There is a risk of adverse events associated with all vaccines and there can be some risks associated with vaccine administration and blood collection procedures like pain, redness, itch, swelling, fever, feverishness, chills, joint pains, muscle pains, fatigue, headache, malaise, nausea, vomiting, diarrhea etc. However, in most cases the adverse events are mild and self-limiting but can require medication and/or hospitalization in rare cases. Participants suffering from any adverse event causally related to the to the trial intervention will be facilitated and the cost of treatment including laboratory investigations will be provided to them. The participants will also be compensated for their time, the inconvenience of getting jabs and providing blood samples.

Confidentiality of all the data collected from the population is a top priority. All the names and personal information regarding any individual will not to be disclosed separately. The data will be published collectively. All the names present in the forms will be de linked and forms will be coded accordingly all the data files will be password protected. Data that will be shared with University of Oxford, International Vaccine Institute (IVI), Seoul, Republic of Korea, Ragon Institute, Harvard School of Medicine, USA, National Institute of Health (NIH) Pakistan will have multi-layered security with several layers of encryption to protect data. Blood samples from patients enrolled will be stored at our research office in Infectious disease research laboratory at Aga Khan University Karachi, labelled with identification numbers not participant name. During the storage, only dedicated members of our study team will have access to the samples. De-identified research data maybe be stored indefinitely. If volunteers consent to be contacted for future research, a record of this consent will be recorded, retained, and stored securely and separately from the research data. If volunteers consent to have their samples stored and used for future research, information about their consent form will be retained and stored securely as per Biobanking procedures and SOPs. Identifiable information such as contact details will be stored for a minimum of 5 years from the end of the study. This includes storage of consent forms. Storage of data will be reviewed every 5 years and files will be confidentially destroyed if storage is no longer required. During the storage, only the local PIs and researchers designated by them will have access to the data or samples.

ELIGIBILITY:
Inclusion Criteria:

- Adult male and female volunteers aged 18 years and above and volunteers with well controlled mild or moderate comorbidities will be enrolled to participate in trial.

* Participant is willing and able to give written informed consent for participation in the trial.
* Male or Female aged 18 years or above and in good health as determined by a trial clinician. Participants may have well controlled mild-moderate comorbidity.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Residing in the study areas.

Exclusion Criteria:

The participant may not enter in the trial if ANY of the following apply:

* Pregnant women or those who are planning to conceive within next 70 days.
* Women who are breast feeding
* Already received any COVID-19 vaccine or any other vaccine likely to impact on interpretation of the trial data (e.g., Adenovirus vectored vaccines).
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient state; asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting ≤14 days)
* History of allergic disease or reactions likely to be exacerbated by any component of study vaccines (e.g., hypersensitivity to the active substance of the COVID-19 vaccines included in the study groups
* Any history of anaphylaxis.
* Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* Bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder), or prior history of thrombotic events and/or significant bleeding or bruising following IM injections or venipuncture.
* Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e., warfarin)
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness (mild/moderate well controlled comorbidities are allowed)
* History of active or previous auto-immune neurological disorders (e.g., multiple sclerosis, Guillain-Barre syndrome, transverse myelitis). Bell's palsy will not be an exclusion criterion.
* History of laboratory confirmed COVID-19 within 6 months prior to enrolment (history of SARS-CoV-2 detection by PCR or antibody to SARS-CoV-2).
* Scheduled elective surgery during the trial.
* Participants enrolled in any other research trial.
* Participants planning to migrate out of the study area within 2 years of the study.

Temporary Exclusion Criteria:

If the volunteer has any of the following, they will not be enrolled that day.

* Acute respiratory illness (moderate or severe illness with or without fever)
* Fever (temperature greater than 38°C) They may be considered for enrolment later in the trial if they recover in sufficient time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | At weeks 14 and 38
  Anti-spike IgG antibodies by ELISA will be measured in serum

SECONDARY OUTCOMES:
Secondary Endpoint 1a | Through study completion, an average of 2 and a half years
  Serious adverse events (SAE) and adverse events of special interest (AESI) assessed through phone calls using a structured questionnaire
Secondary Endpoint 1b | Within 7 days post each dose
  Solicited local and systemic reactions assessed through phone calls using a structured questionnaire
Secondary Endpoint 1c | Within 28 days post each dose
  Unsolicited adverse reactions assessed through phone calls using a structured questionnaire
Secondary Endpoint 1d | Up to 3 months post booster dose
  Medically attended adverse reactions assessed through phone calls using a structured questionnaire
Secondary Endpoint 1e:1 | From baseline to 4 weeks post each dose
  Detect changes in urea levels in serum Unit of measurement: mg/dL
Secondary Endpoint 1e:2 | From baseline to 4 weeks post each dose
  Detect changes in sodium levels in serum Unit of measurement: mEq/L
Secondary Endpoint 1e:3 | From baseline to 4 weeks post each dose
  Detect changes in potassium levels in serum Unit of measurement: mEq/L
Secondary Endpoint 1e:4 | From baseline to 4 weeks post each dose
  Detect changes in creatinine levels in serum Unit of measurement: mg/dL
Secondary Endpoint 1e:5 | From baseline to 4 weeks post each dose
  Detect changes in bilirubin levels in serum Unit of measurement: mg/dL
Secondary Endpoint 1e:6 | From baseline to 4 weeks post each dose
  Detect changes in Alanine Aminotransferase (ALT) levels in serum Unit of measurement: IU/L
Secondary Endpoint 1e:7 | From baseline to 4 weeks post each dose
  Detect changes in ALT-phosphatase levels in serum Unit of measurement: IU/L
Secondary Endpoint 1e:8 | From baseline to 4 weeks post each dose
  Detect changes in albumin levels in serum Unit of measurement: g/dL
Secondary Endpoint 1e:9 | From baseline to 4 weeks post each dose
  Detect changes in Aspartate Aminotransferase (AST) levels in serum Unit of measurement: units/L
Secondary Endpoint 1e:10 | From baseline to 4 weeks post each dose
  Detect changes in blood hematology tests through complete blood count (CBC) using whole blood
Secondary Endpoint 2 | At day 0, and weeks 4, 14, 24, 28, 48, 60 and 96 as per schedule of events (only immunology cohort) and at baseline and 4 weeks post booster dose in general cohort
  Neutralizing antibody response (pseudo-virus neutralization assay) against SARS-CoV-2 in serum
Secondary Endpoint 3a | Measured at Day 0, and Weeks 4, 10, 14, 24, 28, 48, 60 and 96 as per schedule of events (in full cohort)
  Anti-spike IgG responses measured by ELISA will be measured in serum
Secondary Endpoint 3b | Measured at Day 0, and Week 2, 14, 24, 48, 60, and 96 as per schedule of events (in full cohort)
  Anti-nucleocapsid IgG will be measured in serum
Secondary Endpoint 3c | At Day 0, and week 2, 4, 10, 12, 14, 24, 48, 96 (immunology cohort)
  ELISpot assays will be performed using peripheral blood mononuclear cells polymorphonuclear cells (PBMC)

OTHER OUTCOMES:
Exploratory Endpoint 1a | Within 1 week of breakthrough infection among the participants
  Neutralizing antibody response (pseudo-virus neutralization assay) against SARS-CoV-2 and anti-spike IgG responses measured by ELISA in serum
Exploratory Endpoint 1b | Througout the study
  Sequencing of SARS-CoV-2 viruses of breakthrough infections in vaccine recipients by extracting DNA from nasal swabs
Exploratory Endpoint 1c | Througout the study
  NNeutralizing antibody response (pseudo-virus neutralization assay) against SARS-CoV-2 VOCs circulating in Pakistan in serum through ELISAVOCs circulating in Pakistan
Exploratory Endpoint 1d | Througout the study
  Intracellular cytokine staining (ICS) will be performed to assess the phenotypic characteristics of CD4 and CD8 T cells recognizing the antigen by high throughput multicolor flow cytometry by extracting peripheral blood mononuclear cells (PBMC)
Exploratory Endpoint 1e | Througout the study
  Strategic stage-gated Systems Serology analysis using Luminex in serum samples

CONTACTS AND LOCATIONS:
Overall Officials: Farah Qamar, Principal Investigator — Aga Khan University Hospital, Pakistan (AKU); Tahir Yousafzai, Study Director — Aga Khan University Hospital, Pakistan (AKU); Zahra Hassan, Study Director — Aga Khan University Hospital, Pakistan (AKU); Junaid Iqbal, Study Director — Aga Khan University Hospital, Pakistan (AKU); Kiran Iqbal, Study Director — Aga Khan University Hospital, Pakistan (AKU); Sonia Qureshi, Study Director — Aga Khan University Hospital, Pakistan (AKU); Maria Fletcher, Study Director — Aga Khan University Hospital, Pakistan (AKU); Najeeha Iqbal, Study Director — Aga Khan University Hospital, Pakistan (AKU); Momin Kazi, Study Director — Aga Khan University Hospital, Pakistan (AKU); Shazia Sultana, Study Director — Aga Khan University Hospital, Pakistan (AKU); Andrew Pollard, Study Director — University of Oxford; Matthew Snape, Study Director — University of Oxford; Teresa Lambe, Study Director — University of Oxford; Xinxue Liu, Study Director — University of Oxford; Anh Wartel, Study Director — International Vaccine Institute (IVI), Korea; Jean-Louis Excler, Study Director — International Vaccine Institute (IVI), Korea; Deok-Ryun Kim, Study Director — International Vaccine Institute (IVI), Korea; Galit Alter, Study Director — Ragon Institute, Harvard School of Medicine, USA; Aamir Ikram, Study Director — National Institute of Health (NIH) Pakistan; Ghazala Parveen, Study Director — National Institute of Health (NIH) Pakistan; Firdous Nawaz Khan, Study Director — National Institute of Health (NIH) Pakistan; Omera Naseer, Study Director — National Institute of Health (NIH) Pakistan
Locations (3):
- Pakistan (3):
  - National Institute of Health, Islamabad, Punjab Province
  - Chughtai Lab, Lahore, Punjab Province
  - Aga Khan University, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawat K, Kumari P, Saha L. COVID-19 vaccine: A recent update in pipeline vaccines, their design and development strategies. Eur J Pharmacol. 2021 Feb 5;892:173751. doi: 10.1016/j.ejphar.2020.173751. Epub 2020 Nov 25. PMID 33245898
- [Background] Dai L, Gao GF. Viral targets for vaccines against COVID-19. Nat Rev Immunol. 2021 Feb;21(2):73-82. doi: 10.1038/s41577-020-00480-0. Epub 2020 Dec 18. PMID 33340022
- [Background] Kahn JS, McIntosh K. History and recent advances in coronavirus discovery. Pediatr Infect Dis J. 2005 Nov;24(11 Suppl):S223-7, discussion S226. doi: 10.1097/01.inf.0000188166.17324.60. PMID 16378050
- [Background] Cui J, Li F, Shi ZL. Origin and evolution of pathogenic coronaviruses. Nat Rev Microbiol. 2019 Mar;17(3):181-192. doi: 10.1038/s41579-018-0118-9. PMID 30531947
- [Background] Perlman S. Another Decade, Another Coronavirus. N Engl J Med. 2020 Feb 20;382(8):760-762. doi: 10.1056/NEJMe2001126. Epub 2020 Jan 24. No abstract available. PMID 31978944
- [Background] Shang J, Wan Y, Liu C, Yount B, Gully K, Yang Y, Auerbach A, Peng G, Baric R, Li F. Structure of mouse coronavirus spike protein complexed with receptor reveals mechanism for viral entry. PLoS Pathog. 2020 Mar 9;16(3):e1008392. doi: 10.1371/journal.ppat.1008392. eCollection 2020 Mar. PMID 32150576
- [Background] Seyed Hosseini E, Riahi Kashani N, Nikzad H, Azadbakht J, Hassani Bafrani H, Haddad Kashani H. The novel coronavirus Disease-2019 (COVID-19): Mechanism of action, detection and recent therapeutic strategies. Virology. 2020 Dec;551:1-9. doi: 10.1016/j.virol.2020.08.011. Epub 2020 Sep 24. PMID 33010669
- [Background] Cheng VC, Wong SC, Chuang VW, So SY, Chen JH, Sridhar S, To KK, Chan JF, Hung IF, Ho PL, Yuen KY. The role of community-wide wearing of face mask for control of coronavirus disease 2019 (COVID-19) epidemic due to SARS-CoV-2. J Infect. 2020 Jul;81(1):107-114. doi: 10.1016/j.jinf.2020.04.024. Epub 2020 Apr 23. PMID 32335167
- [Background] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Background] Rizwana S SZ. Second Wave of COVID-19 Pandemic: Its deleterious and mortal repercussion in Pakistan. Journal of Rawalpindi Medical College. 2020;24(4):288-9.
- [Background] DRAP. Emergency use authorization of COVID-19 vaccines by DRAP. 2021.
- [Background] DAWN. Govt okays Russian vaccine for 'emergency use'. 2021.
- [Background] DAWN. Chinese CanSinoBio becomes fourth Covid-19 vaccine to be approved for emergency use in Pakistan. 2021.
- [Background] Google News: Vaccine dose overview. 2021.
- [Background] David W. Kimberlin M, FAAP; Michael T. Brady, MD, FAAP; Mary Anne Jackson, MD, FAAP; Sarah S. Long, MD, FAAP. Red Book Report of the Committee on Infectious Diseases. 31st Edition ed2018-2021.
- [Background] Masood T. Factors affecting full immunization coverage among children aged 12-23 months in urban and rural areas of Sindh. Indian Journal of Science and Technology. 2020;13:1283-92.
- [Background] SAMAA. COVID-19 vaccine updates in Pakistan and around the world. 2021.
- [Background] NPR. Pakistan's Vaccine Worries: Rich People And Conspiracy Theorists. 2021.
- [Background] Dagotto G, Yu J, Barouch DH. Approaches and Challenges in SARS-CoV-2 Vaccine Development. Cell Host Microbe. 2020 Sep 9;28(3):364-370. doi: 10.1016/j.chom.2020.08.002. Epub 2020 Aug 10. PMID 32798444
- [Background] Dolzhikova IV, Zubkova OV, Tukhvatulin AI, Dzharullaeva AS, Tukhvatulina NM, Shcheblyakov DV, Shmarov MM, Tokarskaya EA, Simakova YV, Egorova DA, Scherbinin DN, Tutykhina IL, Lysenko AA, Kostarnoy AV, Gancheva PG, Ozharovskaya TA, Belugin BV, Kolobukhina LV, Pantyukhov VB, Syromyatnikova SI, Shatokhina IV, Sizikova TV, Rumyantseva IG, Andrus AF, Boyarskaya NV, Voytyuk AN, Babira VF, Volchikhina SV, Kutaev DA, Bel'skih AN, Zhdanov KV, Zakharenko SM, Borisevich SV, Logunov DY, Naroditsky BS, Gintsburg AL. Safety and immunogenicity of GamEvac-Combi, a heterologous VSV- and Ad5-vectored Ebola vaccine: An open phase I/II trial in healthy adults in Russia. Hum Vaccin Immunother. 2017 Mar 4;13(3):613-620. doi: 10.1080/21645515.2016.1238535. Epub 2017 Feb 2. PMID 28152326
- [Background] Lu S. Heterologous prime-boost vaccination. Curr Opin Immunol. 2009 Jun;21(3):346-51. doi: 10.1016/j.coi.2009.05.016. Epub 2009 Jun 6. PMID 19500964
- [Background] Excler JL, Kim JH. Novel prime-boost vaccine strategies against HIV-1. Expert Rev Vaccines. 2019 Aug;18(8):765-779. doi: 10.1080/14760584.2019.1640117. Epub 2019 Jul 9. PMID 31271322
- [Background] He Q, Mao Q, An C, Zhang J, Gao F, Bian L, Li C, Liang Z, Xu M, Wang J. Heterologous prime-boost: breaking the protective immune response bottleneck of COVID-19 vaccine candidates. Emerg Microbes Infect. 2021 Dec;10(1):629-637. doi: 10.1080/22221751.2021.1902245. PMID 33691606
- [Background] Garnett CT, Erdman D, Xu W, Gooding LR. Prevalence and quantitation of species C adenovirus DNA in human mucosal lymphocytes. J Virol. 2002 Nov;76(21):10608-16. doi: 10.1128/jvi.76.21.10608-10616.2002. PMID 12368303
- [Background] Kroger AT, Atkinson WL, Marcuse EK, Pickering LK; Advisory Committee on Immunization Practices (ACIP) Centers for Disease Control and Prevention (CDC). General recommendations on immunization: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2006 Dec 1;55(RR-15):1-48. PMID 17136024
- [Background] Lu LL, Suscovich TJ, Fortune SM, Alter G. Beyond binding: antibody effector functions in infectious diseases. Nat Rev Immunol. 2018 Jan;18(1):46-61. doi: 10.1038/nri.2017.106. Epub 2017 Oct 24. PMID 29063907
- [Background] Coughlin MM, Prabhakar BS. Neutralizing human monoclonal antibodies to severe acute respiratory syndrome coronavirus: target, mechanism of action, and therapeutic potential. Rev Med Virol. 2012 Jan;22(1):2-17. doi: 10.1002/rmv.706. Epub 2011 Sep 8. PMID 21905149
- [Background] Du L, He Y, Zhou Y, Liu S, Zheng BJ, Jiang S. The spike protein of SARS-CoV--a target for vaccine and therapeutic development. Nat Rev Microbiol. 2009 Mar;7(3):226-36. doi: 10.1038/nrmicro2090. Epub 2009 Feb 9. PMID 19198616
- [Background] Chung AW, Kumar MP, Arnold KB, Yu WH, Schoen MK, Dunphy LJ, Suscovich TJ, Frahm N, Linde C, Mahan AE, Hoffner M, Streeck H, Ackerman ME, McElrath MJ, Schuitemaker H, Pau MG, Baden LR, Kim JH, Michael NL, Barouch DH, Lauffenburger DA, Alter G. Dissecting Polyclonal Vaccine-Induced Humoral Immunity against HIV Using Systems Serology. Cell. 2015 Nov 5;163(4):988-98. doi: 10.1016/j.cell.2015.10.027. PMID 26544943
- [Background] Wise J. Covid-19: New data on Oxford AstraZeneca vaccine backs 12 week dosing interval. BMJ. 2021 Feb 3;372:n326. doi: 10.1136/bmj.n326. No abstract available. PMID 33536232
- [Background] REG 174 INFORMATION FOR UK HEALTHCARE PROFESSIONALS. 2021
- [Background] TRTWORLD. Pakistan says CanSinoBIO vaccine 65.7% effective in trials - latest updates. 2021.
- [Background] SAMAA. COVID-19: Pakistan begins vaccinations as deaths reach 11,802. 2021
- [Background] Saleem AF, Mach O, Quadri F, Khan A, Bhatti Z, Rehman NU, Zaidi S, Weldon WC, Oberste SM, Salama M, Sutter RW, Zaidi AK. Immunogenicity of poliovirus vaccines in chronically malnourished infants: a randomized controlled trial in Pakistan. Vaccine. 2015 Jun 4;33(24):2757-63. doi: 10.1016/j.vaccine.2015.04.055. Epub 2015 Apr 24. PMID 25917673
- [Background] Saleem AF, Mach O, Yousafzai MT, Khan A, Weldon WC, Oberste MS, Sutter RW, Zaidi AKM. Needle adapters for intradermal administration of fractional dose of inactivated poliovirus vaccine: Evaluation of immunogenicity and programmatic feasibility in Pakistan. Vaccine. 2017 May 31;35(24):3209-3214. doi: 10.1016/j.vaccine.2017.04.075. Epub 2017 May 4. PMID 28479178
- [Background] Saleem AF, Mach O, Yousafzai MT, Khan A, Weldon WC, Steven Oberste M, Zaidi SS, Alam MM, Quadri F, Sutter RW, Zaidi AKM. Immunogenicity of Different Routine Poliovirus Vaccination Schedules: A Randomized, Controlled Trial in Karachi, Pakistan. J Infect Dis. 2018 Jan 17;217(3):443-450. doi: 10.1093/infdis/jix577. PMID 29126173
- [Background] Saleem AF, Yousafzai MT, Mach O, Khan A, Quadri F, Weldon WC, Oberste MS, Zaidi SS, Alam MM, Sutter RW, Zaidi AKM. Evaluation of vaccine derived poliovirus type 2 outbreak response options: A randomized controlled trial, Karachi, Pakistan. Vaccine. 2018 Mar 20;36(13):1766-1771. doi: 10.1016/j.vaccine.2018.02.051. Epub 2018 Feb 21. PMID 29477307
- [Background] Yousafzai MT, Saleem AF, Mach O, Baig A, Sutter RW, Zaidi AKM. Feasibility of conducting intradermal vaccination campaign with inactivated poliovirus vaccine using Tropis intradermal needle free injection system, Karachi, Pakistan. Heliyon. 2017 Sep 18;3(8):e00395. doi: 10.1016/j.heliyon.2017.e00395. eCollection 2017 Aug. PMID 29333501
- [Background] Saleem AF, Mach O, Yousafzai MT, Kazi Z, Baig A, Sajid M, Jeyaseelan V, Sutter RW, Zaidi AKM. One-Year Decline of Poliovirus Antibodies Following Fractional-Dose Inactivated Poliovirus Vaccine. J Infect Dis. 2021 Apr 8;223(7):1214-1221. doi: 10.1093/infdis/jiaa504. PMID 32798224
- [Background] Riaz A, Mohiuddin S, Husain S, Yousafzai MT, Sajid M, Kabir F, Rehman NU, Mirza W, Salam B, Nadeem N, Pardhan K, Khan KMA, Raza SJ, Arif F, Iqbal K, Zuberi HK, Whitney CG, Omer SB, Zaidi AKM, Ali A; Pakistan Pneumococcal Vaccine Study Group. Effectiveness of 10-valent pneumococcal conjugate vaccine against vaccine-type invasive pneumococcal disease in Pakistan. Int J Infect Dis. 2019 Mar;80:28-33. doi: 10.1016/j.ijid.2018.12.007. Epub 2018 Dec 18. PMID 30576865
- [Background] Qamar FN, Yousafzai MT, Khaliq A, Karim S, Memon H, Junejo A, Baig I, Rahman N, Bhurgry S, Afroz H, Sami U. Adverse events following immunization with typhoid conjugate vaccine in an outbreak setting in Hyderabad, Pakistan. Vaccine. 2020 Apr 23;38(19):3518-3523. doi: 10.1016/j.vaccine.2020.03.028. Epub 2020 Mar 20. PMID 32201138
- [Background] Qamar FN, Batool R, Qureshi S, Ali M, Sadaf T, Mehmood J, Iqbal K, Sultan A, Duff N, Yousafzai MT. Strategies to Improve Coverage of Typhoid Conjugate Vaccine (TCV) Immunization Campaign in Karachi, Pakistan. Vaccines (Basel). 2020 Nov 19;8(4):697. doi: 10.3390/vaccines8040697. PMID 33228111
- See also: Patel D. Poverty in Pakistan: Numerous efforts, many numbers, not enough results 2015 — http://www.aiddata.org/blog/poverty-in-pakistan-numerous-efforts-many-numbers-not-enough-results

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT05162482/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT05162482/ICF_001.pdf